CLINICAL TRIAL: NCT03178669
Title: A Randomised Dose-Optimisation Study to Evaluate the Efficacy and Safety of Cobitolimod in Moderate to Severe Active Ulcerative Colitis Patients
Brief Title: The Efficacy of Cobitolimod in Patients With Moderate to Severe Active Ulcerative Colitis
Acronym: CONDUCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InDex Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSUC-01/16; 2016-004217-26 (EudraCT Number)
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Results first posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Ulcerative Colitis
Keywords: Colitis, Ulcerative; Gastrointestinal Diseases; Inflammatory Bowel Disease; Immunomodulator Therapy; Glucocorticoids; Anti-Inflammatory Agents; Therapeutic uses; Kappaproct; IDX0150; DIMS0150
MeSH Terms: conditions — Colitis, Ulcerative; Gastrointestinal Diseases; Inflammatory Bowel Diseases | interventions — cobitolimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cobitolimod Dose 2x31 mg (Experimental): Dose 31 mg of cobitolimod at 2 occasions, placebo at 2 occasions
  Interventions: Drug: cobitolimod
- Cobitolimod Dose 2x125 mg (Experimental): Dose 125 mg of cobitolimod at 2 occasions, placebo at 2 occasions
  Interventions: Drug: cobitolimod
- Cobitolimod Dose 2x250 mg (Experimental): Dose 250 mg of cobitolimod at 2 occasions, placebo at 2 occasions
  Interventions: Drug: cobitolimod
- Cobitolimod Dose 4x125 mg (Experimental): Dose 125 mg of cobitolimod, at 4 occasions
  Interventions: Drug: cobitolimod
- Placebo (Placebo Comparator): Placebo at four occasions
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: cobitolimod — Rectal administration
  Other Names: Kappaproct
  Arms: Cobitolimod Dose 2x125 mg; Cobitolimod Dose 2x250 mg; Cobitolimod Dose 2x31 mg; Cobitolimod Dose 4x125 mg
Drug: Placebo — Solution manufactured to mimic cobitolimod
  Other Names: Placebo (for cobitolimod)
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate efficacy of cobitolimod treatment at different dose levels and frequencies compared to placebo in patients with moderate to severe left-sided ulcerative colitis.

DETAILED DESCRIPTION:
This was a Phase IIb study in patients with moderate to severe left-sided ulcerative colitis. Patients either received cobitolimod 31 mg, 125 mg or 250 mg at two occasions or 125 mg or placebo at four occasions during a 3-weeks period. To ensure blindness, patients received active treatment at two occasions and placebo at the other two occasions. Blood, stool, and tissue samples was collected at various time points throughout the study to evaluate safety and efficacy. Primary endpoint was evaluated at week 6.

Duration of participation for patients was approximately 12 weeks (from screening to final follow-up visit).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Established diagnosis of Ulcerative Colitis (UC)
* Moderately to severely active left sided UC assessed by central reading
* Current oral 5-Aminosalicylic Acid (5-ASA)/ Sulphasalazine (SP) use or a history of oral 5-ASA/SP use
* Current Glucocorticosteroids (GCS) use or history of GCS dependency, refractory, or intolerance
* Demonstrated an inadequate response, loss of response, or intolerance to at least one of the following agents:

  * Immunomodulators
  * Tumor Necrosis Factor alpha (TNF-α) inhibitors and/or anti-integrins

Exclusion Criteria:

* Suspicion of differential diagnosis
* Acute fulminant UC and/or signs of systemic toxicity
* UC limited to the rectum (disease which extend <15 cm above the anal verge)
* History of malignancy
* History or presence of any clinically significant disorder
* Concomitant treatment with cyclosporine, methotrexate, tacrolimus, TNF-α inhibitors, anti-integrins or similar immunosuppressants and immunomodulators
* Treatment with rectal GCS, 5-ASA/SP or tacrolimus
* Long term treatment with antibiotics or non-steroidal anti-inflammatory drugs (NSAIDs)
* Serious active infection
* Gastrointestinal infections
* Currently receiving parenteral nutrition or blood transfusions
* Females who are lactating or have a positive serum pregnancy test
* Women of childbearing potential not using reliable contraceptive methods
* Concurrent participation in another clinical study
* Previous exposure to cobitolimod

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raja Atreya, Principal Investigator — Friedrich-Alexander University Erlangen-Nuremberg
Locations (64):
- 1, Prague, Czechia
- France (9):
  - 2, Amiens
  - 3, Caen
  - 4, Clichy
  - 5, Grenoble
  - 6, Nice
  - 7, Pierre-Bénite
  - 8, Saint-Etienne
  - 9, Toulouse
  - 10, Vandœuvre-lès-Nancy
- Germany (10):
  - 11, Augsburg
  - 12, Berlin
  - 13, Erlangen
  - 14, Hamburg
  - 15, Hanover
  - 16, Heidelberg
  - 17, Leipzig
  - 18, Lüneburg
  - 19, Mannheim
  - 20, München
- Hungary (5):
  - 22, Békéscsaba
  - 21, Budapest
  - 23, Debrecen
  - 24, Mosonmagyaróvár
  - 25, Pécs
- Poland (10):
  - 26, Częstochowa
  - 27, Krakow
  - 28, Ksawerów
  - 33, Lodz
  - 29, Lublin
  - 30, Poznan
  - 31, Sopot
  - 32, Warsaw
  - 33, Wroclaw
  - 32, Włocławek
- Russia (11):
  - 34, Cheboksary
  - 36, Kazan'
  - 37, Kirov
  - 38, Moscow
  - 39, Novosibirsk
  - 40, Ryazan
  - 41, Saint Petersburg
  - 42, Stavropol
  - 43, Tver'
  - 44, Ufa
  - 35, Yekaterinburg
- 45, Belgrade, Serbia
- Spain (5):
  - 46, Ferrol
  - 47, Fuenlabrada
  - 48, Madrid
  - 49, Seville
  - 50, Valencia
- 51, Uppsala, Sweden
- Ukraine (11):
  - 52, Chernivtsi
  - 53, Dnipro
  - 54, Ivano-Frankivsk
  - 55, Kharkiv
  - 56, Kiev
  - 57, Lutsk
  - 58, Lviv
  - 59, Odesa
  - 60, Sumy
  - 62, Uzhhorod
  - 61, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Atreya R, Peyrin-Biroulet L, Klymenko A, Augustyn M, Bakulin I, Slankamenac D, Miheller P, Gasbarrini A, Hebuterne X, Arnesson K, Knittel T, Kowalski J, Neurath MF, Sandborn WJ, Reinisch W; CONDUCT study group. Cobitolimod for moderate-to-severe, left-sided ulcerative colitis (CONDUCT): a phase 2b randomised, double-blind, placebo-controlled, dose-ranging induction trial. Lancet Gastroenterol Hepatol. 2020 Dec;5(12):1063-1075. doi: 10.1016/S2468-1253(20)30301-0. Epub 2020 Oct 5. PMID 33031757

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 patient in the 2x31 mg and one patient in the 4x125 mg was never treated with study drug and excluded from analysis.
Period: Overall Study
Arm/Group | Cobitolimod Dose 2x31 mg | Cobitolimod Dose 2x125 mg | Cobitolimod Dose 2x250 mg | Cobitolimod Dose 4x125 mg | Placebo
Started | 40 | 43 | 42 | 42 | 44
Completed Week 6 (Completed Week 6) | 35 | 42 | 36 | 38 | 42
Completed (Completed Week 10) | 35 | 42 | 35 | 38 | 40
Not Completed | 5 | 1 | 7 | 4 | 4
Not completed — Adverse Event | 4 | 1 | 4 | 2 | 2
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cobitolimod Dose 2x31 mg | Cobitolimod Dose 2x125 mg | Cobitolimod Dose 2x250 mg | Cobitolimod Dose 4x125 mg | Placebo | Total
Number analyzed (Participants) | 40 | 43 | 42 | 42 | 44 | 211
Age, Customized [Mean (Standard Deviation); unit: years] | 47.4 (16.4) | 47.0 (16.9) | 46.2 (14.0) | 47.2 (14.9) | 45.5 (15.2) | 46.6 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 23 | 16 | 18 | 11 | 82
  Male | 26 | 20 | 26 | 24 | 33 | 129
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity : Asian | 0 | 1 | 1 | 2 | 2 | 6
  Ethnicity : White | 39 | 42 | 40 | 39 | 42 | 202
  Ethnicity : Other | 1 | 0 | 1 | 1 | 0 | 3
Body weight [Mean (Standard Deviation); unit: kg] | 75.5 (16.70) | 71.5 (14.85) | 73.3 (13.15) | 73.1 (17.53) | 78.1 (12.89) | 74.3 (15.14)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.1 (4.54) | 24.7 (4.65) | 24.5 (3.70) | 24.7 (5.06) | 25.9 (4.80) | 25.0 (4.56)
Tobacco use at screening [Count of Participants; unit: Participants]
  Never smoked | 30 | 28 | 30 | 30 | 31 | 149
  Current smoker | 1 | 2 | 2 | 1 | 2 | 8
  Former smoker | 9 | 13 | 10 | 11 | 11 | 54
Total inflammatory Bowel Disease Questionnaire score (IBDQ) [Mean (Standard Deviation); unit: scores on a scale] — The IBDQ is an instrument used to assess quality of life in participants. It includes 32 questions on 4 domains : Bowel Systems (10 items), Emotional Function (12 items), Social Function (5 items), and Systemic Function (5 items). A total IBDQ score is calculated by summing the scores from each domain; the total IBDQ score ranges from 32 to 224, with lower scores reflecting worse health.
  scores on a scale | 131.9 (28.11) | 140.1 (32.46) | 131.5 (36.64) | 120.9 (34.81) | 133.9 (28.58) | 131.7 (32.59)
Duration of Ulcerative Colitis (UC) [Mean (Standard Deviation); unit: years] | 7.88 (6.480) | 8.46 (7.431) | 7.89 (6.830) | 8.14 (6.772) | 7.36 (7.277) | 7.94 (6.920)
Stool frequency per day [Mean (Standard Deviation); unit: Stools per day] | 6.3 (2.93) | 5.0 (1.83) | 5.7 (2.73) | 5.7 (2.56) | 5.9 (3.04) | 5.7 (2.62)
Mayo score [Mean (Standard Deviation); unit: scores on a scale] — The Mayo score is sum of 4 sub-scores (i.e., stool frequency, rectal bleeding, endoscopic findings (excluding friability at grade 1), and physician's global assessment); each rated on a scale from 0 to 3, with higher scores indicating more severe disease. The total Mayo score value ranges from 0 to 12. Higher values represent worse disease.
  scores on a scale | 8.5 (1.2) | 8.0 (1.8) | 8.5 (1.3) | 8.3 (1.7) | 8.3 (1.6) | 8.3 (1.5)
Mayo stool frequency subscore [Count of Participants; unit: Participants] — Mayo stool frequency subscore: 0=normal, 1=one to two stools per day more than normal, 2=three to four stools per day more than normal, 3=more than four stools per day more than normal.
  Participants
    0 | 2 | 8 | 3 | 2 | 4 | 19
    1 | 7 | 11 | 8 | 8 | 10 | 44
    2 | 17 | 10 | 17 | 16 | 10 | 70
    3 | 14 | 14 | 14 | 16 | 20 | 78
Mayo rectal bleeding subscore [Count of Participants; unit: Participants] — Mayo rectal bleeding sub-score: 0=none, 1=visible blood with stool less than half the time, 2=visible blood with stool half the time or more, 3=passing blood alone.
  Participants
    0 | 0 | 4 | 0 | 1 | 4 | 9
    1 | 11 | 9 | 16 | 17 | 15 | 68
    2 | 27 | 26 | 21 | 21 | 22 | 117
    3 | 2 | 4 | 5 | 3 | 3 | 17
Mayo endoscopic subscore [Count of Participants; unit: Participants] — Mayo endoscopic subscore: 2=moderate disease (marked erythema, absent vascular pattern, friability, erosions), 3=severe disease (spontaneous bleeding, ulceration).
  Participants
    2 | 18 | 17 | 17 | 19 | 20 | 91
    3 | 22 | 26 | 25 | 23 | 24 | 120
Mayo Physicians Global Assessment (PGA) subscore [Count of Participants; unit: Participants] — Mayo PGA subscore:1=mild disease, 2=moderate disease, 3=severe disease.
  Participants
    1 | 2 | 4 | 3 | 4 | 3 | 16
    2 | 32 | 34 | 32 | 31 | 31 | 160
    3 | 6 | 5 | 7 | 7 | 10 | 35
Disease extent [Count of Participants; unit: Participants]
  Rectosigmoid | 23 | 22 | 19 | 23 | 21 | 108
  Descending colon | 17 | 21 | 23 | 19 | 23 | 103
Nancy Histological Index (NHI) score [Count of Participants; unit: Participants] — Nancy Histological Index (NHI) classifies histologic status, a score from 0 to 4. Grade 0= no histological findings, grade 1= no acute acute inflammatory infiltrate, grade 2= acute inflammatory cells infiltrate and no ulceration 3= acute inflammatory cells infiltrate and no ulceration 4= ulceration. The most severe observation across all segments is used for the final NHI score. A higher score indicates more severe disease. Population: Missing NHI score for 2 patients
  Participants
    0: number analyzed (Participants) | 40 | 43 | 40 | 42 | 44 | 209
    0 | 0 | 0 | 2 | 0 | 1 | 3
    1: number analyzed (Participants) | 40 | 43 | 40 | 42 | 44 | 209
    1 | 0 | 2 | 0 | 1 | 2 | 5
    2: number analyzed (Participants) | 40 | 43 | 40 | 42 | 44 | 209
    2 | 4 | 4 | 3 | 6 | 3 | 20
    3: number analyzed (Participants) | 40 | 43 | 40 | 42 | 44 | 209
    3 | 14 | 18 | 17 | 14 | 13 | 76
    4: number analyzed (Participants) | 40 | 43 | 40 | 42 | 44 | 209
    4 | 22 | 19 | 18 | 21 | 25 | 105
Faecal calprotectin [Mean (Standard Deviation); unit: mg/kg] | 3563 (6256) | 3389 (5669) | 2654 (4294) | 3730 (4954) | 3263 (5379) | 3313 (5292)
C-reactive protein (CRP) [Mean (Standard Deviation); unit: mg/L] | 7.6 (16.2) | 4.9 (5.0) | 7.1 (9.5) | 9.7 (16.9) | 8.1 (12.1) | 7.5 (11.9)
Concomitant Ulcerative Colitis(UC) medication [Count of Participants; unit: Participants]
  5-aminosalicylic acid (5-ASA) | 35 | 38 | 33 | 33 | 39 | 178
  Corticosteroids | 18 | 13 | 17 | 14 | 17 | 79
  Thiopurines | 9 | 6 | 9 | 10 | 7 | 41
Previous UC therapy [Count of Participants; unit: Participants]
  Thiopurines | 39 | 40 | 42 | 40 | 42 | 203
  Anti-TNF Therapy | 9 | 10 | 9 | 12 | 8 | 48
  Vedolizumab | 4 | 3 | 5 | 3 | 0 | 15
  Tofacitinib | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Remission
Description: Patients with clinical remission at Week 6 (yes=1, no=0), defined by Modified Mayo sub scores, i) rectal bleeding of 0, ii) stool frequency of 0 or 1 (with at least one point decrease from Baseline, Week 0), and iii) endoscopy score of 0 or 1 (excluding friability).
Time Frame: 6 weeks after first treatment
Population: The full analysis set (FAS), was based on the intention-to-treat (ITT) principles, which consists of all randomised patients who meet the inclusion criteria (as assessed by the investigator on the inclusion/exclusion criteria form), and receive at least one dose of the study drug (active or placebo). Missing data was replaced using Non Responder Imputation (NRI). Number of observed data is presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cobitolimod Dose 2x31 mg | Cobitolimod Dose 2x125 mg | Cobitolimod Dose 2x250 mg | Cobitolimod Dose 4x125 mg | Placebo
Number analyzed (Participants) | 40 | 43 | 42 | 42 | 44
Participants | 5 | 2 | 9 | 4 | 3
Statistical Analysis 1: Comparison: Cobitolimod Dose 2x31 mg vs Placebo; Test type: Superiority; p = 0.1806, Cochran-Mantel-Haenszel — one-sided and adjusted for stratification factors, p values of less than 0.10 were regarded as statistically significant; Odds Ratio (OR) = 2.0, 80% CI 2-sided [0.75 to 5.47]
Statistical Analysis 2: Comparison: Cobitolimod Dose 2x125 mg vs Placebo; Test type: Superiority; p = 0.6649, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.7, 80% CI 2-sided [0.20 to 2.24]
Statistical Analysis 3: Comparison: Cobitolimod Dose 2x250 mg vs Placebo; Test type: Superiority; p = 0.0247, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.8, 80% CI 2-sided [1.53 to 9.47]
Statistical Analysis 4: Comparison: Cobitolimod Dose 4x125 mg vs Placebo; Test type: Superiority; p = 0.3279, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.4, 80% CI 2-sided [0.52 to 3.88]

2. Secondary Outcome: Modified Clinical Remission
Description: Patients with modified clinical remission at Week 6 (yes=1, no=0), defined by the Modified Mayo score ≤ 2 and sub scores, i) rectal bleeding of 0, ii) stool frequency of 0 or 1 (with at least one point decrease from Baseline, Week 0), iii) endoscopy score of 0 or 1 (excluding friability ) and iiii) physician´s global assessment (PGA) of 0 or 1
Time Frame: Week 6
Population: The full analysis set (FAS), was based on the intention-to-treat (ITT) principles, which consists of all randomised patients who meet the inclusion criteria (as assessed by the investigator on the inclusion/exclusion criteria form), and receive at least one dose of the study drug (active or placebo). Missing data was replaced using Placebo Multiple Imputation (PMI). Number of observed data is presented in the table.
Measure: Count of Participants; unit: Participants
Arm/Group | Cobitolimod Dose 2x31 mg | Cobitolimod Dose 2x125 mg | Cobitolimod Dose 2x250 mg | Cobitolimod Dose 4x125 mg | Placebo
Number analyzed (Participants) | 33 | 41 | 35 | 39 | 39
Participants | 5 | 1 | 7 | 3 | 3
Statistical Analysis 1: Comparison: Cobitolimod Dose 2x31 mg vs Placebo; Test type: Superiority; p = 0.2115, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.9, 80% CI 2-sided [0.69 to 4.99]
Statistical Analysis 2: Comparison: Cobitolimod Dose 2x125 mg vs Placebo; Test type: Superiority; p = 0.8498, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.3, 80% CI 2-sided [0.06 to 1.34]
Statistical Analysis 3: Comparison: Cobitolimod Dose 2x250 mg vs Placebo; Test type: Superiority; p = 0.0977, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.6, 80% CI 2-sided [1.01 to 6.62]
Statistical Analysis 4: Comparison: Cobitolimod Dose 4x125 mg vs Placebo; Test type: Superiority; p = 0.5220, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.0, 80% CI 2-sided [0.32 to 2.84]

3. Secondary Outcome: Symptomatic Remission
Description: Patients with symptomatic remission at Week 6 (yes=1, no=0), defined by the Mayo sub scores, i) rectal bleeding of 0, ii) stool frequency of 0 or 1 (with at least one point decrease from Baseline, Week 0), (patient reported outcome)
Time Frame: Week 6
Population: The full analysis set (FAS), was based on the intention-to-treat (ITT) principles, which consists of all randomised patients who meet the inclusion criteria (as assessed by the investigator on the inclusion/exclusion criteria form), and receive at least one dose of the study drug (active or placebo). Missing data was replaced using Placebo Multiple Imputation (PMI). Number of observed data is presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cobitolimod Dose 2x31 mg | Cobitolimod Dose 2x125 mg | Cobitolimod Dose 2x250 mg | Cobitolimod Dose 4x125 mg | Placebo
Number analyzed (Participants) | 37 | 42 | 37 | 40 | 43
Participants | 10 | 11 | 13 | 10 | 9
Statistical Analysis 1: Comparison: Cobitolimod Dose 2x31 mg vs Placebo; Test type: Superiority; p = 0.2335, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.5, 80% CI 2-sided [0.74 to 2.94]
Statistical Analysis 2: Comparison: Cobitolimod Dose 2x125 mg vs Placebo; Test type: Superiority; p = 0.2511, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.4, 80% CI 2-sided [0.73 to 2.69]
Statistical Analysis 3: Comparison: Cobitolimod Dose 2x250 mg vs Placebo; Test type: Superiority; p = 0.1162, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.8, 80% CI 2-sided [0.96 to 3.52]
Statistical Analysis 4: Comparison: Cobitolimod Dose 4x125 mg vs Placebo; Test type: Superiority; p = 0.3467, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.2, 80% CI 2-sided [0.63 to 2.40]

4. Secondary Outcome: Clinical Response
Description: Patients with clinical response at Week 6 (yes=1, no=0), defined as clinical remission or a three point and ≥30 % decrease from Baseline, Week 0 in the sum of the Modified Mayo score, i) rectal bleeding, ii) stool frequency and iii) endoscopy score (excluding friability), iiii) physicians global assessment (PGA)
Time Frame: Week 6
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cobitolimod Dose 2x31 mg | Cobitolimod Dose 2x125 mg | Cobitolimod Dose 2x250 mg | Cobitolimod Dose 4x125 mg | Placebo
Number analyzed (Participants) | 33 | 41 | 35 | 39 | 39
Participants | 17 | 18 | 20 | 15 | 20
Statistical Analysis 1: Comparison: Cobitolimod Dose 2x31 mg vs Placebo; Test type: Superiority; p = 0.6326, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.9, 80% CI 2-sided [0.50 to 1.50]
Statistical Analysis 2: Comparison: Cobitolimod Dose 2x125 mg vs Placebo; Test type: Superiority; p = 0.7127, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.8, 80% CI 2-sided [0.45 to 1.37]
Statistical Analysis 3: Comparison: Cobitolimod Dose 2x250 mg vs Placebo; Test type: Superiority; p = 0.2658, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.3, 80% CI 2-sided [0.75 to 2.34]
Statistical Analysis 4: Comparison: Cobitolimod Dose 4x125 mg vs Placebo; Test type: Superiority; p = 0.8301, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.6, 80% CI 2-sided [0.36 to 1.16]

5. Secondary Outcome: Endoscopic Remission
Description: Patients with endoscopic remission at Week 6 (yes=1, no=0), defined by the Modified Mayo endoscopic sub score of 0 or 1 (excluding friability)
Time Frame: Week 6
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cobitolimod Dose 2x31 mg | Cobitolimod Dose 2x125 mg | Cobitolimod Dose 2x250 mg | Cobitolimod Dose 4x125 mg | Placebo
Number analyzed (Participants) | 34 | 41 | 37 | 39 | 40
Participants | 7 | 5 | 15 | 10 | 12
Statistical Analysis 1: Comparison: Cobitolimod Dose 2x31 mg vs Placebo; Test type: Superiority; p = 0.7994, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.6, 80% CI 2-sided [0.32 to 1.27]
Statistical Analysis 2: Comparison: Cobitolimod Dose 2x125 mg vs Placebo; Test type: Superiority; p = 0.9665, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.3, 80% CI 2-sided [0.16 to 0.72]
Statistical Analysis 3: Comparison: Cobitolimod Dose 2x250 mg vs Placebo; Test type: Superiority; p = 0.2049, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.5, 80% CI 2-sided [0.80 to 2.82]
Statistical Analysis 4: Comparison: Cobitolimod Dose 4x125 mg vs Placebo; Test type: Superiority; p = 0.6504, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.8, 80% CI 2-sided [0.42 to 1.60]

6. Secondary Outcome: Histological Remission
Description: Patients with histological remission at Week 6 (yes=1, no=0), defined by the Nancy histological index of grade 0 or 1
Time Frame: Week 6
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cobitolimod Dose 2x31 mg | Cobitolimod Dose 2x125 mg | Cobitolimod Dose 2x250 mg | Cobitolimod Dose 4x125 mg | Placebo
Number analyzed (Participants) | 35 | 41 | 37 | 39 | 41
Participants | 4 | 5 | 8 | 7 | 10
Statistical Analysis 1: Comparison: Cobitolimod Dose 2x31 mg vs Placebo; Test type: Superiority; p = 0.9207, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.4, 80% CI 2-sided [0.18 to 0.93]
Statistical Analysis 2: Comparison: Cobitolimod Dose 2x125 mg vs Placebo; Test type: Superiority; p = 0.9228, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.4, 80% CI 2-sided [0.19 to 0.92]
Statistical Analysis 3: Comparison: Cobitolimod Dose 2x250 mg vs Placebo; Test type: Superiority; p = 0.6636, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.8, 80% CI 2-sided [0.39 to 1.61]
Statistical Analysis 4: Comparison: Cobitolimod Dose 4x125 mg vs Placebo; Test type: Superiority; p = 0.7449, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.7, 80% CI 2-sided [0.34 to 1.41]

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) was collected from the date of signed informed consent. During the screening period up to first treatment only AEs related to a study specific procedures should be reported. AEs were reported up to follow up visit at Week 10 (from first treatment)
Arm/Group | Cobitolimod Dose 2x31 mg | Cobitolimod Dose 2x125 mg | Cobitolimod Dose 2x250 mg | Cobitolimod Dose 4x125 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/43 | 0/42 | 0/42 | 1/44
Serious Adverse Events (participants affected / at risk) | 2/40 | 0/43 | 4/42 | 2/42 | 2/44
Other Adverse Events (participants affected / at risk) | 5/40 | 12/43 | 8/42 | 10/42 | 11/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cobitolimod Dose 2x31 mg (N=40) | Cobitolimod Dose 2x125 mg (N=43) | Cobitolimod Dose 2x250 mg (N=42) | Cobitolimod Dose 4x125 mg (N=42) | Placebo (N=44)
Ulcerative colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cobitolimod Dose 2x31 mg (N=40) | Cobitolimod Dose 2x125 mg (N=43) | Cobitolimod Dose 2x250 mg (N=42) | Cobitolimod Dose 4x125 mg (N=42) | Placebo (N=44)
Ulcerative colitis (Gastrointestinal disorders) | 2 (3) | 5 (5) | 4 (5) | 2 (3) | 3 (4)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (4)
Viral upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 5 (5) | 2 (2) | 2 (4) | 0 (0)
Faecal calprotectin increased (Investigations) | 2 (2) | 0 (0) | 0 | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT03178669/Prot_SAP_000.pdf